CLINICAL TRIAL: NCT01821248
Title: A Multicenter Phase II Trial of Preoperative Chemotherapy With Gemcitabine/ Cisplatin /S-1 (GCS) for Biliary Tract Cancers With Lymph Node Metastasis Diagnosed by Fluorodeoxyglucose Positron Emission Tomography (FDG-PET)
Brief Title: A Phase II Trial of Preoperative Chemotherapy for Biliary Tract Cancer (BTC) With Node Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1201; UMIN000009831 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-03-22; First posted 2013-03-29 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Cisplatin, S-1 (Experimental): 1000mg/m2/day1, 25mg/m2/day1, 100mg/body/day1-7
  Interventions: Drug: Gemcitabine, Cisplatin, S-1

INTERVENTIONS:
Drug: Gemcitabine, Cisplatin, S-1 — Preoperative chemotherapy (GCS) 3 cycles -FDG-PET- surgery
  GCS therapy Gemcitabine 1000mg/m2/day1 Cisplatin 25mg/m2/day1 S-1 100mg/body/day1-7
  Other Names: Gemcitabine；gemzer; Cisplatin；Cispulan; S-1；TS-1

SUMMARY:
To evaluate the efficacy and the safety of preoperative chemotherapy with Gemcitabine/ Cisplatin /S-1 for biliary tract cancers with lymph node metastasis by FDG-PET.

DETAILED DESCRIPTION:
Biliary tract cancer is one of the most lethal malignancies worldwide, with surgery representing the only potentially curative treatment for this disease. However, many patients are diagnosed as far advanced stage, which is too late for curative resection, and even if surgery can be performed, the likelihood of relapse is very high. Lymph node metastasis is the most powerful prognostic factor in biliary tract cancer, which makes accurate preoperative assessment of lymph node metastasis important for indication of resection. However, the diagnostic accuracy, sensitivity, and specificity of conventional imaging techniques, including computed tomography (CT) and magnetic resonance imaging (MRI), seem to be insufficient for accurate detection of lymph node metastasis. Previously, the investigators reported FDG-PET is useful for prediction of lymph node metastasis.

On the other hand, gemcitabine has been widely used to treat the patients with unresectable or recurrent biliary tract cancer. In the Advanced Biliary tract Cancer (ABC)-02 study, the first prospective multicenter phase III study in this field, the combination of gemcitabine/cisplatin was compared with gemcitabine monotherapy and found that the combination regimen significantly prolonged Median Survival Time (MST) (from 8.1 to 11.7 months; P < 0.001). Gemcitabine/cisplatin combination therapy is now considered to be the standard regimen for advanced biliary tract cancer. S-1 is an oral fluoropyrimidine prodrug that has confirmed efficacy against various solid tumors, both alone and in combination with other cytotoxic drugs. S-1 monotherapy has yielded good results against advanced biliary tract cancer and gemcitabine/S-1 combination therapy has yielded promising results with acceptable toxicity levels for patients with advanced biliary tract cancer.

Furthermore, the investigators reported the safety and efficacy of adding S-1 to gemcitabine/cisplatin combination regimen (GCS) for advanced biliary tract cancer.

In this study, the investigators evaluate the efficacy and the safety of preoperative chemotherapy with Gemcitabine/ Cisplatin /S-1 for biliary tract cancers with lymph node metastasis by FDG-PET

ELIGIBILITY:
Inclusion Criteria:

1. Patients with radiologically proven biliary tract cancer.
2. No extra-hepatic disease.
3. No prior therapy.
4. The function of the liver is kept as satisfied after hepatectomy.
5. No chronic liver damage.
6. Patients of age over 20 years.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
8. Sufficient organ function (neutrophil count >=1,500/mm3 and platelet count >=100,000/mm3, Hemoglobin >=9.0g/dL, Aspartate transaminase (AST)/alanine aminotransferase (ALT) <=150 IU/L, total bilirubin <=1.5 mg/dL , creatinine <=1.2 mg/dL , creatinine clearance >=60 mL/min) 9.Patients obtained written informed consent.

Exclusion Criteria:

1. Massive abdominal effusion requiring treatment.
2. Active concomitant malignancy.
3. The case suspected of infection.
4. Patients with water solubility diarrhea.
5. Mental disease or psychotic manifestation.
6. Under continuous steroid therapy.
7. Patients with acute myocardial infarction.
8. Patients with severe complications.
9. Pregnancy or the desire to preserve fecundity.
10. Serious drug hypersensitivity or a history of drug allergy.
11. Any patients judged by the investigator to be unfit to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-07-23 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Curative resection rate | 14weeks
  The primary endpoint is designated to evaluate curative resection rate after preoperative chemotherapy with GCS for Biliary Tract Cancers with lymph node metastasis diagnosed by FDG-PET.

SECONDARY OUTCOMES:
Response rate and toxicity | 10 weeks
  Secondary endpoints include response rate according to FDG-PET and the incidence of adverse events evaluated by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Etsuro Hatano, MD, PhD, Study Director — Kyoto University
Locations (1):
- Kyoto University Hospital, Kyoto, Japan